

## EMPHASIS-lung ETOP 3-12

A randomized phase III trial of erlotinib versus docetaxel in patients with advanced squamous cell non-small cell lung cancer who failed first line platinumbased doublet chemotherapy stratified by VeriStrat Good vs VeriStrat Poor

E r l o t i n o h a s i g n a t u r e i n o n - s m a l l u n g c a n c e r

## A clinical trial of ETOP

## NCT01652469

| SAP VERSION | V.1 |
|-----------------------------|-----------------------------|
| SAP VERSION DATE | 07.01.2015 |
| TRIAL STATISTICIAN | Urania Dafni |
| TRIAL PRIMARY INVESTIGATORS | Egbert Smit, Solange Peters |
| DSMB SAP AUTHOR | Marie Kassapian |



Figure 1: Patient flowchart



Figure 2a: expected vs observed accrual



Figure 2b: Cumulative accrual by treatment arm



**Figure 3:** Time on follow-up by treatment arm (N=xxx)



**Figure 4:** Time on treatment by treatment arm (N=xxx)



Figure 5a: Distribution of adverse events



Figure 5b: Distribution of adverse events by treatment arm



Figure 6a: Distribution of serious adverse events



Figure 6b: Distribution of serious adverse events by treatment arm



Figure 7a: Distribution of serious adverse events



Figure 7b: Distribution of serious adverse events by treatment arm



Figure 8a: Distribution of serious adverse events according to CTCAE Version 4



Figure 8b: Distribution of serious adverse events by treatment arm according to CTCAE Version 4



Figure 9a: Severity of adverse events



Figure 9b: Severity of adverse events by treatment arm



Figure 10a: Severity of adverse events according to CTCAE Version 4



 $\textbf{\textit{Figure 10b:} Severity of adverse events by treatment arm according to \textit{CTCAE Version 4}}$ 



Figure 11a: Maximum severity of adverse event per patient



Figure 11b: Maximum severity of adverse event per patient by treatment arm



Figure 12a: Distribution of adverse events



Figure 12b: Distribution of adverse events by treatment arm



Figure 13a: Distribution of adverse events according to CTCAE Version 4



Figure 13b: Distribution of adverse events by treatment arm according to CTCAE Version 4



Figure 14: Progression-free Survival (N=xxx)



**Figure 15:** Progression-free Survival by VeriStrat status (N=xxx)



Figure 16: Overall Survival (N=xxx)



Figure 17: Overall Survival by VeriStrat status (N=xxx)